CLINICAL TRIAL: NCT06169137
Title: Pilot Study of Isocaloric Time Restricted Eating on Ketone Metabolism and Immunoregulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10001746; 001746-DK
Record Dates: First submitted 2023-12-11; First posted 2023-12-13 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08-20

CONDITIONS: Obesity; Body Weight
Keywords: Diet; Time Restricted Eating; Inflammation; Ketone Bodies
MeSH Terms: conditions — Obesity; Body Weight; Intermittent Fasting; Inflammation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Premenopausal women (lean and obese) (Experimental): Ages 18-50 yearsBMI 18.0-24.5 mg/k^2 or BMI > 30 mg/k^2
  Interventions: Behavioral: Early Time-Restricted Eating; Behavioral: Conventional dietary regimen (12-hr, 9:30a-9:30p)

INTERVENTIONS:
Behavioral: Early Time-Restricted Eating — Participants will be provided all meals to consume within a 6-hour timeframe (9:30-3:30p)
Behavioral: Conventional dietary regimen (12-hr, 9:30a-9:30p) — Participants will be provided all meals to consume within a 12-hour timeframe (9:30a-9:30p)

SUMMARY:
Background:

Time restricted eating (TRE) is a form of fasting in which a person eats only during a set window of time, which is usually between 4 and 10 hours each day. Researchers want to know more about how TRE may affect health.

Objective:

To learn how TRE affects women with different body sizes.

Eligibility:

Healthy women aged 18 to 50 years.

Design:

Participants will have 2 visits: 1 screening visit and one 5-day stay in the clinic.

Participants will fast before both visits. They will have a physical exam with blood tests. They will talk to a nutritionist about the foods they eat. They will lay under a clear hood for up to 45 minutes during a test that measures how many calories they burn while resting.

Participants will keep a food diary for up to 7 days before their clinic stay. They will apply a continuous glucose monitor the day before they go to the clinic. This is a device that attaches to the skin of the stomach. They will wear this device throughout their clinic stay.

All meals will be provided during the clinic stay. Participants will follow TRE on 3 days. They will answer survey questions and have tests during their stay, including:

* DXA (dual energy X-ray absorptiometry) scan. Participants will lie on a padded table. Their body will be scanned to measure how much muscle, bone, fat, and other tissues they have.
* Stable isotope tracer study. Small amounts of sugar and other substances will be given through a tube attached to a needle inserted into a vein in the arm. Blood samples will be collected.

DETAILED DESCRIPTION:
Study Description:

Intermittent fasting confers anti-inflammatory effects, although underlying metabolic mechanisms are poorly defined. This pilot study will explore ketone bodies as a mediator of inflammation in response to time restricted eating (TRE-6-hr feeding/18-hr fast) without caloric restriction compared to a more conventional dietary regimen (12-hr feeding/12-hr fast) in women classified as obese and lean.

Objectives:

Primary Aim 1: Quantify ketone body (beta-OHB) whole-body turnover after short-term early 6-hr TRE compared to a conventional 12-hr dietary regimen in women.

Primary Aim 2: Quantify CD4+ T cell responses after short-term early 6-hr TRE compared to a conventional 12-hr dietary regimen in women.

Secondary Aim 1: Determine metabolic response to short-term early 6-hr TRE in lean women vs women with obesity.

Secondary Aim 2: Determine immunomodulatory effects of short-term early 6-hr TRE in lean women vs women with obesity.

Exploratory Aim 1: Evaluate ketone body, hormonal, and cardiometabolic responses after short-term early 6-hr TRE compared to a conventional 12-hr dietary regimen in women classified as lean and with obesity.

Exploratory Aim 2: Evaluate effects of short-term early 6-hr TRE on perceived appetite, stress, and gastrointestinal symptoms.

Endpoints:

Primary:

1. Change from admission day 0 in ketone body (beta-OHB) rate of appearance (Ra) after three days of 6-hr TRE
2. Change from admission in CD4+ T cell responsiveness (Th17 polarization) after three days of 6-hr TRE

Secondary:

1. Change from admission day 0 in post-absorptive glucose Ra quantified using [6,6-2H2]glucose (intravenous) after three days 6- hr TRE
2. Change from admission day 0 in ketone body Ra in lean vs. obese women after three days 6-hr TRE
3. CD4+ T cell responsiveness (Th17 polarization) in lean vs. obese women after three days 6-hr TRE
4. Evaluation of ketone biology in isolated CD4+ T cells, using biochemical analysis and analysis of metabolic reprograming at the gene regulatory level

Exploratory:

1. Circulating ketone body concentrations at admission day 0 and after 3 days of TRE
2. Hormonal mediators of metabolic status (morning cortisol, fasting insulin and glucagon/incretins, thyroid hormones, sex hormone binding globulin, anti-mullerian hormone)
3. Cardiometabolic biomarkers (glycemic, lipid, and inflammatory; trimethylamine N-oxide [TMAO])
4. Perceived appetite, stress, and gastrointestinal symptom scores

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study
2. Women between ages 18-50 years who are premenopausal (defined as regular menses and/or FSH <ULN)
3. BMI of 18-24.9 or >=30 kg/m^2
4. In good general health as evidenced by medical history and/or screening laboratory evaluation.
5. Agreement to adhere to Lifestyle Considerations throughout study duration

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Diagnosis/treatment for immune/inflammatory disorder or other metabolic conditions that would interfere with study parameters, including diabetes, chronic kidney, chronic liver disease, history of hypoglycemia, and thyroid disease (with the exception of chronic controlled hypothyroidism as measured by TSH within normal limits)
2. Current use of antihyperglycemic medications, systemic steroids, adrenergic-stimulating agents, or medications affecting sleep, circadian rhythms, or metabolism which affect parameters under investigation (examples include oral contraceptives, anti-diabetic agents, nicotinamide riboside, tryptophan, vitamin B3 supplements)
3. Caffeine consumption in excess of approximately 300 mg (approximately three 8-oz cups of coffee) daily
4. Factors that affect circadian rhythms including individuals who perform overnight shift work, report irregular sleep and/or eating schedules, and who regularly fast for more than 15 hours/day
5. History of an eating disorder by self-report or medical history
6. Food allergies/intolerances or dietary patterns that would prohibit consumption of metabolic diet
7. Inability to provide informed consent
8. Pregnancy or lactation
9. Unstable weight with more than 5% body weight change in last previous 3 months
10. Engaged in competitive sports training and/ or unwilling to comply with exercise regimen in this protocol.
11. Consumption of more than 3 servings of alcohol daily
12. Current smoker or regular tobacco use, vaping, or other forms of nicotine within prior 3 months

This study will recruit only women. The study design was informed by our Protocol NCT04728165 which investigates an identical 6:18h TRE intervention in males who are healthy and those with psoriasis. Based on our pilot data in men, the current study is needed to test our hypothesis in women. This study in women is a critical next step to replicate the findings in women and to understand sex-specific differences in TRE response and ketone metabolism.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2027-02-05 (Estimated); Study Completion 2027-02-05 (Estimated)

PRIMARY OUTCOMES:
Change in ketone body (beta hydroxybutyrate) rate of appearance (Ra) | Day 0, Day 3
  Within subject difference in ketone body (beta hydroxybutyrate) rate of appearance (Ra) after 3 days of 6-hr TRE compared to a 12-hr eating window regimen
Change in CD4+ T cell responsiveness (Th17 polarization) | Day 0, Day 3
  Within subject difference in CD4+ T cell response after 3 days of 6-hr TRE compared to a 12-hr eating window regimen

SECONDARY OUTCOMES:
Change in post-absorptive glucose rate of appearance (Ra) | Day 0, Day 3
  Within subjective difference in glucose Ra quantified using [6,6- 2H2]glucose (intravenous) after 3 days of 6-hr TRE compared to a 12-hr eating window regimen
Change in ketone body rate of appearance (Ra) in lean women vs women with obesity | Day 0, Day 3
  Between subject comparison in ketone body rate of appearance after 3 days of 6-hr TRE compared to a 12-hr eating window regimen in lean women vs women with obesity
Change in CD4+ T cell responsiveness (Th17 polarization) in lean women vs women with obesity | Day 0, Day 3
  Between subject comparison in CD4+ T cell response after 3 days of 6-hr TRE compared to a 12-hr eating window regimen in lean women vs women with obesity
Ketone biology in isolated CD4+ T cells | Day 0, Day 3
  Biochemical and metabolic reprogramming analysis at the gene regulatory level

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie T Chung, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will provide raw data (without identifying information) to journals or other researchers upon request.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be provided upon request within 1 year after publication and will be available to indefinitely
Access Criteria: The PI will accept requests from other researchers who are examining pertinent outcomes

REFERENCES:
- [Background] Han K, Nguyen A, Traba J, Yao X, Kaler M, Huffstutler RD, Levine SJ, Sack MN. A Pilot Study To Investigate the Immune-Modulatory Effects of Fasting in Steroid-Naive Mild Asthmatics. J Immunol. 2018 Sep 1;201(5):1382-1388. doi: 10.4049/jimmunol.1800585. Epub 2018 Jul 18. PMID 30021766
- [Background] Puchalska P, Crawford PA. Metabolic and Signaling Roles of Ketone Bodies in Health and Disease. Annu Rev Nutr. 2021 Oct 11;41:49-77. doi: 10.1146/annurev-nutr-111120-111518. PMID 34633859
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001746-DK.html